CLINICAL TRIAL: NCT05042570
Title: The Effect of Instrument Assisted Soft Tissue Mobilization and Stretching Exercises on Flexibility, Spasticity and Balance in Individuals With Cerebral Palsy
Brief Title: The Effect of Instrument Assisted Soft Tissue Mobilization and Stretching Exercises in Cerebral Palsy
Acronym: IASTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eren Avcıl, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EAvcil2
Record Dates: First submitted 2021-08-01; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Instrument Assisted Soft Tissue Mobilization; Stretching Exercises
MeSH Terms: conditions — Cerebral Palsy | interventions — Muscle Stretching Exercises; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instrument Assisted Soft Tissue Mobilization (Experimental): Group 1 (n=13): Each session will consist of 40 minutes. An additional 10 minutes of IASTM will be performed to the 30-minute NDT program.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Stretching Exercises (Experimental): Group 2 (n=13): Each session will consist of 40 minutes. In addition to the NDT program applied for 30 minutes, 10 minutes of Stretching Exercises will be performed.
  Interventions: Other: Stretching Exercises
- Control (Active Comparator): Group 3 (n=13): Each session will consist of 40 minutes. There will be no additional application to the NDT program, which is applied for 40 minutes, and it will be included as a control group in the study.
  Interventions: Other: Control Group / NDT program

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — * This technique will be performed using instruments of different sizes, shapes and treatment styles.
  * During the application, instruments will be applied to loosen the muscle tissue and fascia by gliding on the tissue at certain angles.
  * The muscle groups to be treated with IASTM are gastrocnemius, soleus and tibialis posterior. It will also be applied to the superficial and deep fascia.
  * The instrument will be sterilized before treatment.
  * IASTM treatment will be applied without damaging the tissue after massaging cream is applied to the muscle fibers with the instrument.
  Arms: Instrument Assisted Soft Tissue Mobilization
Other: Stretching Exercises — * The muscle groups to be applied stretching exercises are gastrocinemius, soleus and tibialis posterior. It will also be applied to the superficial and deep fascia.
  * 3 different functional stretching exercises will be applied;
  * With the hands supported on the wall and with the help of the physiotherapist, the affected extremity is behind the knee in full extension m. gastrocnemius stretching exercise,
  * With the hands supported on the wall and with the help of the physiotherapist, the knee is partially flexed, with the affected extremity behind. soleus stretching exercise,
  * It is a stretching exercise that will be applied by asking the patient to squat without lifting his heels, with the patient's hands supported by the physiotherapist.
  Arms: Stretching Exercises
Other: Control Group / NDT program — * Efforts to eliminate tone disorders,
  * Sensory-perception-motor integrity development studies,
  * Activities aimed at facilitating movements in daily life,
  * Stretching and strengthening exercises due to muscle shortness and weakness,
  * Studies to increase lower and upper extremity functionality,
  * It will include the training of activities such as standing up, walking and balance.
  Arms: Control

SUMMARY:
The aim of the study; To investigate the effects of Instrument Assisted Soft Tissue Mobilizations and Stretching Exercises on flexibility, spasticity, balance and functional mobility in patients with CP.

DETAILED DESCRIPTION:
Various intervention studies; reported positive results with EDYDM after carpal tunnel syndrome, myofascial trigger point, chronic low back pain, nonspecific thoracic spine pain, ankle instability, mastectomy and total joint arthroplasty. Observational studies have shown positive results in improving posterior shoulder range of motion, hip, knee, and ankle ROM.

There is no study in the literature with EDYDM in patients with CP. Many of the problems in which EDDM is applied for fascia and muscle mobilization in different diseases are also seen in patients with CP. In current rehabilitation methods, Stretching Exercises are applied for muscle and fascia shortening. The advantages of the applications over each other are unknown. Our study is planned as a study with high original value as it is the first study to be conducted using EDYDM in cases with CP. In our study, the effectiveness of EDYDM treatment, which will increase the effectiveness of stretching exercises in CP or can be an alternative treatment approach in cases with CP, will be compared with Stretching Exercises.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Unilateral Spastic Type Cerebral Palsy by the health committee report,
* Level I or II according to GMFCS,
* Being between the ages of 5-18,
* No Botulinum Toxin (Botox) injection in the last 6 months,
* Not using any medication that may affect muscle tone,
* Passive ankle dorsiflexion + 10o and passive plantar flexion -25o,
* Families and children agree to participate voluntarily in the study.

Exclusion Criteria:

* Having undergone any lower extremity surgery,
* Tone in plantar flexors is level IV according to MAS,
* Presence of advanced contracture in the ankle,
* Presence of any diagnosed cardiac or orthopedic disorder that may prevent the application of the treatment,
* Hearing or vision problems,
* Having a history of epileptic attacks,
* Not having the ability to adapt to exercises (cases with the phrase "Mental Retarde" according to the health report).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | one month
  In the evaluation of the presence of spasticity in patients with CP, the ankle plantar flexors will be based. It is recorded as an assessment of the resistance encountered while passively moving the limb at full range of motion. It is scored as 0, 1, 1+, 2, 3, 4. A value of 0 is the best score without muscle tone increase, while a value of 4 is when the extremity is in a rigid position. Modified Ashworth Scale (MAS) will be used to evaluate spasticity.
Pediatric Berg Balance Scale (PBBS) | one month
  The Pediatric Berg Balance Scale, which is the version of the Berg Balance Scale designed for children by Franjoine et al., will be used to evaluate their functional balance in activities of daily living. The scale consists of 14 sections and each section is scored between 0-4; The highest score that can be obtained from the scale is 56.
Selective Motor Control Test (SMCT) | one month
  Ankle dorsiflexion Selective Motor Control Test will be used in the evaluation of selective movements. This test evaluates the isolated dorsiflexion movement of the ankle and is evaluated between 0-4 according to the selectivity of the ankle dorsiflexion movement in the long sitting position.
Weight-Bearing Lunge Testi (WBLT) | one month
  In order to measure the weight-bearing dorsiflexion ROM, the Weight-Bearing Lunge Test, which is positioned with support from the wall in the closed chain position, will be applied. An increase in ankle dorsiflexion angle will be considered as a positive result.

CONTACTS AND LOCATIONS:
Overall Officials: İpek Yeldan, Prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)